CLINICAL TRIAL: NCT00663780
Title: Pharmacogenomic Analysis of Blood Samples to Identify Polymorphisms That Segregate Responders From Non-Responders Following Treatment With Juvidex of Split Skin Donor Sites in Renovo's Clinical Study RN1004-0082
Brief Title: Pharmacogenomic Analysis of Samples From Subjects in Study RN1004-0082
Status: Completed | Type: Observational
Sponsor: Renovo (Industry)
Responsible Party: Dr Jim Bush, Renovo
Other Study IDs: RN1004-0084
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Last update posted 2009-01-06 (Estimated); Status verified 2009-01

CONDITIONS: Wound
Keywords: pharmacogenomics; polymorphisms; wound healing
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma retained until samples analysed then destroyed
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the study is to identify variations in subjects genetic makeup that segregate responders from non-responders in respect of response to Juvidex in the clinical trial RN1004-0082

DETAILED DESCRIPTION:
Injury to the skin results in the physical disruption of the normal cellular architecture and triggers wound healing: a process involving inflammation, cell proliferation and migration, cell recruitment, angiogenesis and extracellular matrix deposition. Growth factors and cytokines released from inflammatory cells dictate the function of those cells present within the wound. There is a clinical need for treatments that accelerate healing, as current therapies in this field are largely based on empirical treatments and are often ineffective or inadequate.Juvidex contains as an active ingredient mannose-6-phosphate (M-6-P), a naturally occurring low molecular weight monosaccharide. The proposed mechanism of action for Juvidex is antagonistic and involves inhibiting the activation of TGF-β1 and TGF-β2. Juvidex is being developed by Renovo as a therapeutic agent administered to accelerate the healing of acute wounds.

Technological advances in genetics are providing scientists with the tools necessary to investigate the relationships between genetic variation and unmanipulated and drug-influenced wound healing outcomes such as the speed of healing. Determining the link between genetic variation and drug response (pharmacogenomics) is becoming an increasingly important part of drug development. For example, Iressa, which antagonises the tyrosine kinase activity of the epithelial growth factor receptor (EGFR) only works in people that have a specific variation (or polymorphism) in the DNA sequence of the EGFR gene. For Renovo, comparing the genetic make-up - (genotypes) - of subjects who respond well and those who respond poorly to a treatment, as well as those who naturally heal faster or whose wounds heal more slowly, may help to better define the most appropriate group of patients in which to target a given treatment. An additional benefit of exploring genotypes in well-defined patient populations will be to help to improve our understanding of the underlying biology of wound healing and provide new targets for drug discovery and development.

Pharmacogenomics may ultimately lead to improved treatment of wound healing by using more effective drugs and safer prescribing regimes. In order to realise these benefits we need to be able to collect samples for genotyping analysis from the associated clinical trial. Renovo wishes to examine the DNA sequence of patients enrolled into its clinical studies in order to examine the variation in patients capacity to heal wounds. This study will analyse samples from subjects participating in clinical study RN1004-0082, a double blind, placebo controlled trial to investigate the efficacy and safety of two concentrations of Juvidex in accelerating the healing of split thickness skin graft donor sites using different dosing regimes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-85 years who have given written informed consent.
* Subjects have given written informed consent to participate in the study RN1004-0082.

Exclusion Criteria:

* Subjects who are not participating in the study RN1004-0082.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will analyse samples from subjects participating in clinical study RN1004-0082, a double blind, placebo controlled trial to investigate the efficacy and safety of two concentrations of Juvidex in accelerating the healing of split thickness skin graft donor sites using different dosing regimes.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To identify polymorphisms that segregate responders from non-responders in respect of response to Juvidex in the clinical trial RN1004-0082 | Single blood sample

SECONDARY OUTCOMES:
Identify polymorphisms associated with differential healing rates and associate data with additional ongoing clinical studies. | Single Blood Sample

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MBChB. MRCS, Principal Investigator — General Medical Council
Locations (1):
- Clinical Trials Unit, Renovo Limited, Manchester, United Kingdom